CLINICAL TRIAL: NCT04457713
Title: Off-label Use of Anti-cancer Drugs in Norway -a Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut Halvor Bjøro Smeland, Chief Attending Physician, Oslo University Hospital
Other Study IDs: Off Label Study protocol
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Off Label Use
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Off-label drug use, where a marketed drug is used outside its approved indication, may allow early access to new and promising treatments. However, its use can be a source of controversy, due to limited evidence for clinical benefit and lack of cost/QALY-estimates, leading to challenging prioritization issues. The number of drugs suitable for off-label use is expected to further increase in the coming years, owing to the rapid progress in the field of oncology, in particular with the current era of precision medicine and targeted therapies. This also challenges the traditional method of running clinical trials, with eligible patient populations commonly being small, underpinning the importance of gaining supplementary real-world evidence from well performed observational studies.

This prospective observational study will therefore assess real-world outcomes of patients treated with off-label anti-cancer drugs, including efficacy in terms of response rates, time to progression/relapse measures and survival; patient-reported outcome measures (PROMS) and self-reported side-effects/toxicity; as well as collecting blood samples for a biobank for further translational research. Further, the study will give a descriptive analysis of the current practice of off-label use of anti-cancer drugs in Norway, including prevalence estimation and health care related cost analyses.

ELIGIBILITY:
Inclusion Criteria:

* Verified cancer diagnosis (based on radiological, histological/cytological or operative evidence).
* Treatment with off-label anti-cancer drug.
* Age ≥ 18 years
* Able to provide written informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient accepted by the leadership in the Department of Oncology at OUH to receive anti-cancer treatment off-label from the date of start of the study is eligible for inclusion. Of note, this does not include off-label use of drugs used for supportive care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS). | Assessed up to 2 years after end of inclusion
  Time from date of inclusion until the date of first documented progression or date of death from any cause, whichever come first, according to RECIST v1.1
Patients questionnaire EORTC QLQ-C30 | Assessed from inclusion until 2 years after end of treatment
  Assessment of patients reported quality of life, as measured by EORTC QLC30

SECONDARY OUTCOMES:
Objective tumor response rate (ORR) | Assed through study completion, an average of 1 year
  Defined as the proportion of patients with an objective tumor response (either partial response [PR] or complete response [CR] using RECIST v1.1) response (DR), time to next treatment and overall survival (OS)
Duration of response (DR) | Assed through study completion, an average of 1 year
  Duration of response among patients with an objective response, according to RECIST v1.1
Time to next treatment (TTNT) | Assed through study completion, an average of 1 year
  Time from inclusion to institution og next therapy
Overall survival (OS) | Assessed up to 2 years after end of inclusion
  Time from date of inclusion until the date of death from any cause
Fatigue | From inclusion until 2 years after end of treatment
  Assessment of patient reported outcomes, as measured by the Chalder Fatigue Questionnaire (FQ)
Depression | From inclusion until 2 years after end of treatment
  Assessment of patient reported outcomes, as measured by the patient health questionnaire (PHQ-9)
Pain intensity | From inclusion until 2 years after end of treatment
  Assessment of patient reported outcomes, as measured by an 11 point Numerical Rating Scale (NRS) for pain intensity
Adverse event | From inclusion until 2 years after end of treatment
  Patients files and self-report. Classified according to CTCAE v 5.0 and MedDRA
Quality adjusted life years (QALYs) | From inclusion until 2 years after end of treatment
  Patient self reported EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Knut Smeland, PhD/MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway